CLINICAL TRIAL: NCT03247231
Title: Effectiveness and Safety of the Endoscopic Band Ligation Without Resection of ≤15-mm Subepithelial Tumours of the Digestive Tract: a Multicenter Prospective Study
Brief Title: Banding Without Resection in Small Subepithelial Tumours
Acronym: BANDING-SET
Status: Terminated | Type: Observational
Why Stopped: Due to SARS-CoV2 (Covid-19) pandemia
Sponsor: Joan B Gornals (Other)
Responsible Party: Sponsor-Investigator, Joan B Gornals, Principal investigator, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: BANDING-SET
Record Dates: First submitted 2017-03-29; First posted 2017-08-11 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Gastrointestinal Subepithelial Tumors
Keywords: Endoscopic ultrasound; Small gastrointestinal subepithelial tumours; Endoscopic band ligation without resection; Single-incision needle-knife biopsy; Pre-cancerous tumours; Multicenter observational cohort study
MeSH Terms: interventions — Electrosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Endoscopic band ligation without resection — Endoscopic treatment of subepithelial tumors: autoamputation by endoscopic band ligation without resection.
  Other Names: Endoscopic ligation; Endoscopic band ligation without electrosurgery; Band ligation with a mucosectomy device without resection
Procedure: SINK — To obtain sample tissue biopsies after the endoscopic band ligation without resection, performing a single-incision with a needle-knife.
  Other Names: Single-incision needle-knife; Single-incision needle-knife and use of a biopsy forceps device

SUMMARY:
To analyse the effectiveness and safety of endoscopic band ligation without resection in small gastrointestinal subepithelial tumours.

DETAILED DESCRIPTION:
Multicenter prospective study analysing the effectiveness and safety of endoscopic band ligation without resection in small (≤15-mm) gastrointestinal subepithelial tumours.

This endoscopic technique will be complemented with a SINK (single-incision needle-knife) biopsy for ensuring the pathological diagnosis of the treated subepithelial tumour.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age between 18 and 80 years old.
* Endoscopic ultrasound (EUS) image of a gastrointestinal subepithelial tumour (SET) ≤15-mm.
* Patient capable of understanding and signing informed consent form.
* Patient understanding the type of study and complying with the follow-up of complementary tests during the study duration.

EXCLUSION CRITERIA:

* SETs >15-mm.
* SETs with clear diagnosis of EUS benign semiology: ie., lipoma, ectopic pancreas.
* Patients with multiple SETs (e.g., carcinoids).
* Vascular SETs (Doppler effect by EUS).
* Severe coagulation disorder: INR >1.5 not correctible with administration of plasma and/or platelets <50,000/mm3.
* Conditions that preclude upper digestive endoscopy, such as stenosis.
* Pregnancy or breast-feeding.
* Failure to sign informed consent form.
* Patients with functional diversity who are unable to understand the nature and possible consequences of the study, unless there is a competent legal representative.
* Patients unable to adhere to subsequent follow-up requirements.
* Patients with a life expectancy of less than 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subepithelial lesions (SEL) in the gastrointestinal tract.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Removal of the subepithelial tumour (initial clinical success). | 4-6 weeks
  Complete removal and disappearance of the subepithelial tumour at 4-6 weeks by endoscopic ultrasonography control.

SECONDARY OUTCOMES:
Removal of the subepithelial tumour (global clinical success). | 1 year
  Complete removal and disappearance of the subepithelial tumour at 1 year by endoscopic ultrasonography control.
Number of participants with treatment-related adverse events as assessed by American Society of Gastrointestinal Endoscopy (ASGE) guideline. | 1 year
  Incidence of treatment-emergent adverse events, graded by American Society of Gastrointestinal Endoscopy (ASGE) guideline (Ref: Cooton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, et al. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc 2010;71:446-54).
Technical success. | First day
  Correct application of elastic banding.
SINK biopsy efectiveness. | 4-6 weeks
  Positive definitve pathological result rate of single-incision needle-knife (SINK) biopsies permorfed in subeptihelial tumours ligated.
Long-term recurrence. | 5 years
  Recurrence of indeterminate or pre-malignant subepithelial tumours rate at 5 years by endoscopic ultrasonography control.

CONTACTS AND LOCATIONS:
Overall Officials: Joan B Gornals, MD, PhD, Principal Investigator — Endoscopy Unit; Digestive Diseases Department; H. Universitari de Bellvitge.; Francesc Bas-Cutrina, MD, Principal Investigator — Endoscopy Unit; Digestive Diseases Department; H. Universitari de Bellvitge.
Locations (7):
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol (Can Ruti), Badalona, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Catalonia
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona, Catalonia
  - Hospital de Sant Pau i de la Santa Creu, Barcelona, Catalonia
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Catalonia
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida, Catalonia
  - Hospital Universitari Joan XXIII de Tarragona, Tarragona, Catalonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bas-Cutrina F, Consiglieri CF, Bosch-Schips J, Gornals JB. Endoscopic band ligation plus single-incision needle knife biopsy for small subepithelial deep-layer tumor: easy and effective. Endoscopy. 2019 Jul;51(7):E191-E192. doi: 10.1055/a-0875-3958. Epub 2019 Apr 12. No abstract available. PMID 30978731
- [Background] Standards of Practice Committee; Faulx AL, Kothari S, Acosta RD, Agrawal D, Bruining DH, Chandrasekhara V, Eloubeidi MA, Fanelli RD, Gurudu SR, Khashab MA, Lightdale JR, Muthusamy VR, Shaukat A, Qumseya BJ, Wang A, Wani SB, Yang J, DeWitt JM. The role of endoscopy in subepithelial lesions of the GI tract. Gastrointest Endosc. 2017 Jun;85(6):1117-1132. doi: 10.1016/j.gie.2017.02.022. Epub 2017 Apr 3. No abstract available. PMID 28385194
- [Background] ASGE Technology Committee; Hwang JH, Konda V, Abu Dayyeh BK, Chauhan SS, Enestvedt BK, Fujii-Lau LL, Komanduri S, Maple JT, Murad FM, Pannala R, Thosani NC, Banerjee S. Endoscopic mucosal resection. Gastrointest Endosc. 2015 Aug;82(2):215-26. doi: 10.1016/j.gie.2015.05.001. Epub 2015 Jun 12. PMID 26077453
- [Background] Song JH, Kim SG, Chung SJ, Kang HY, Yang SY, Kim YS. Risk of progression for incidental small subepithelial tumors in the upper gastrointestinal tract. Endoscopy. 2015 Aug;47(8):675-9. doi: 10.1055/s-0034-1391967. Epub 2015 May 11. PMID 25961444
- [Background] de la Serna-Higuera C, Perez-Miranda M, Diez-Redondo P, Gil-Simon P, Herranz T, Perez-Martin E, Ochoa C, Caro-Paton A. EUS-guided single-incision needle-knife biopsy: description and results of a new method for tissue sampling of subepithelial GI tumors (with video). Gastrointest Endosc. 2011 Sep;74(3):672-6. doi: 10.1016/j.gie.2011.05.042. PMID 21872716
- [Background] Binmoeller KF, Shah JN, Bhat YM, Kane SD. Suck-ligate-unroof-biopsy by using a detachable 20-mm loop for the diagnosis and therapy of small subepithelial tumors (with video). Gastrointest Endosc. 2014 May;79(5):750-5. doi: 10.1016/j.gie.2013.09.028. Epub 2013 Nov 12. PMID 24238309
- [Background] Ibanez-Sanz G, Gornals JB, Rivas L, Salord S, Paules MJ, Botargues JM, Galan M. Endoscopic band ligation without resection in selected patients for small and superficial upper gastrointestinal tract lesions. Rev Esp Enferm Dig. 2016 May;108(5):250-6. doi: 10.17235/reed.2016.4031/2015. PMID 27022723
- [Background] Bas-Cutrina F, Ballester-Clau R, Gonzalez-Huix F, Gornals JB. Gastric perforation during ligation-assisted endoscopic mucosal resection of a neuroendocrine tumor: banding without resection may be a safer option. Endoscopy. 2020 Oct;52(10):E370-E371. doi: 10.1055/a-1134-4742. Epub 2020 Mar 27. No abstract available. PMID 32219785
- [Derived] Bas-Cutrina F, Loras C, Pardo A, Ballester-Clau R, Huertas C, Guarner-Argente C, Colan-Hernandez J, Consiglieri CF, Andujar X, Vilanova-Serra M, Gonzalez-Huix F, Pardo-Grau L, Maisterra S, Ruiz-Ramirez P, Garcia-Sumalla A, Tebe C, Videla S, Gornals JB. Management of small subepithelial tumors by endoscopic banding without resection and single-incision needle-knife-assisted biopsy sampling: a prospective multicenter study. Gastrointest Endosc. 2023 Dec;98(6):911-921.e8. doi: 10.1016/j.gie.2023.05.057. Epub 2023 May 30. PMID 37263361